CLINICAL TRIAL: NCT05580562
Title: ONC201 for the Treatment of Newly Diagnosed H3 K27M-mutant Diffuse Glioma Following Completion of Radiotherapy: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study
Brief Title: ONC201 in H3 K27M-mutant Diffuse Glioma Following Radiotherapy (the ACTION Study)
Acronym: ACTION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ONC201-108
Expanded Access: NCT04617002 (Approved for marketing)
Record Dates: First submitted 2022-09-27; First posted 2022-10-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: H3 K27M; Glioma
Keywords: H3 K27M; H3 K28M; H3 K27-altered; histone; H3F3A; HIST1H3B; HIST1H3C; H3.1; H3.3; DMG; thalamus; thalamic; midline
MeSH Terms: conditions — Glioma | interventions — TIC10 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ONC201 Twice Weekly Group (Experimental)
  Interventions: Drug: Dordaviprone (ONC201)
- ONC201 Once Weekly Group (Experimental)
  Interventions: Drug: Dordaviprone (ONC201) + Placebo
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dordaviprone (ONC201) — Participants ≥ 52.5 kg will receive 625 mg of ONC201 (5 × 125-mg capsules) dosing days; participants < 52.5 kg will receive a dose (and corresponding number of capsules) scaled by body weight and rounded to 125-mg increments.
  Arms: ONC201 Twice Weekly Group
Drug: Dordaviprone (ONC201) + Placebo — Participants ≥ 52.5 kg will receive 625 mg of ONC201 (5 × 125-mg capsules) or matching placebo on dosing days; participants < 52.5 kg will receive a dose (and corresponding number of capsules) scaled by body weight and rounded to 125-mg increments
  Arms: ONC201 Once Weekly Group
Other: Placebo — Participants will receive placebo (same number of capsules as the ONC201 dose) on dosing days
  Arms: Placebo Group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, international, Phase 3 study in patients with newly diagnosed H3 K27M-mutant diffuse glioma to assess whether treatment with ONC201 following frontline radiotherapy will extend overall survival and progression-free survival in this population. Eligible participants will have histologically diagnosed H3 K27M-mutant diffuse glioma and have completed standard frontline radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study procedures and agree to participate in the study by providing written informed consent (by participant or legally authorized representative), and assent when applicable.
2. Body weight ≥ 10 kg at time of randomization.
3. Histologically diagnosed H3 K27M-mutant diffuse glioma (new diagnosis). Detection of a missense K27M mutation in any histone H3-encoding gene detected by testing of tumor tissue (immunohistochemistry [IHC] or next-generation sequencing [NGS] in a Clinical Laboratory Improvement Amendments [CLIA]-certified or equivalent laboratory). [Site to provide (as available): ≥ 10 unstained formalin-fixed paraffin-embedded (FFPE) slides from tumor tissue.]
4. At least one, high-quality, contrast-enhanced MRI of the brain obtained prior to starting radiotherapy for submission to sponsor's imaging vendor for central read. For participants who had a surgical resection, this scan must be post-resection; for participants who did not have a resection, this scan may be pre- or post-biopsy.
5. At least one, high-quality, contrast-enhanced MRI of the brain obtained 2 to 6 weeks after completion of frontline radiotherapy. If unable to obtain contrast-enhanced imaging due to lack of venous access after multiple attempts, a patient may still be eligible after collection of a nonenhanced MRI of the brain. [Site to also provide all available MRIs completed prior to initiating treatment with study intervention.]
6. Received frontline radiotherapy

   1. Initiated radiotherapy within 12 weeks from the initial diagnosis of H3 K27M-mutant diffuse glioma.
   2. Completed radiotherapy within 2 to 6 weeks prior to randomization
   3. Completed standard fractionated radiotherapy (eg. 54 to 60 Gy in 28 to 33 fractions given over approximately 6 weeks or hypofractionated radiotherapy (eg. 40 Gy in 15 fractions given over approximately 3 weeks).
7. Karnofsky Performance Status or Lansky Performance Status ≥ 70 at time of randomization.
8. Stable or decreasing dose of corticosteroids and anti-seizure medications for 7 days prior to randomization, if applicable. Stable steroid dose is defined as ≤ 2 mg/day increase (based on dexamethasone dose or equivalent dose of an alternative steroid).

Exclusion Criteria:

1. Primary spinal tumor.
2. Diffuse intrinsic pontine glioma (DIPG), defined as tumors with a pontine epicenter and diffuse involvement of the pons.
3. Evidence of leptomeningeal spread of disease or cerebrospinal fluid dissemination.
4. Any known concurrent malignancy.
5. New lesion(s) outside of the radiation field.
6. Received whole-brain radiotherapy.
7. Received proton therapy for glioma.
8. Use of any of the following treatments within the specified time periods prior to randomization:

   1. ONC201 or ONC206 at any time.
   2. Systemic bevacizumab (includes biosimilars) at any time since the initial diagnosis of H3 K27M-mutant diffuse glioma.
   3. Temozolomide within past 3 weeks.
   4. Tumor treating fields at any time.
   5. DRD2 antagonist within past 2 weeks.
   6. Any investigational therapy within past 4 weeks.
   7. Strong CYP3A4 inhibitors within 3 days.
   8. Strong CYP3A4 inducers (includes enzyme-inducing antiepileptic drugs) within 2 weeks.
9. Laboratory test results meeting any of the following parameters within 2 weeks prior to randomization:

   1. Absolute neutrophil count < 1.0 × 109/L or platelets < 75 × 109/L.
   2. Total bilirubin > 1.5 × upper limit of normal (ULN) (participants with Gilbert's syndrome may be included with total bilirubin > 1.5 × ULN if direct bilirubin is ≤ 1.5 × ULN).
   3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN.
   4. Creatinine clearance ≤ 60 mL/min as calculated by the Cockcroft Gault equation (or estimated glomerular filtration rate < 60 mL/min/1.73 m2).
10. QTc > 480 msec (based on mean from triplicate electrocardiograms) during screening.
11. Known hypersensitivity to any excipients used in the study intervention formulation.
12. Pregnant, breastfeeding, or planning to become pregnant while receiving study intervention or within 3 months after the last dose. Participants of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study intervention.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy or psychiatric illness/social situations that would limit compliance with study requirements.
14. Any other condition (eg, medical, psychiatric, or social) that, in the opinion of the investigator, may interfere with participant safety or the ability to complete the study according to the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until date of death from any cause, assessed up to approximately 44 months
  Overall Survival is defined as the time from randomization to death due to any cause.
Progression free survival (PFS) as assessed by using RANO-HGG criteria | From date of randomization until the date of first documented progression assessed up to approximately 44 months
  PFS is defined as time from randomization to disease progression (PD) or death.

SECONDARY OUTCOMES:
Incidence of adverse events | From date of randomization up to 44 months
  Incidence of overall, treatment-related, Grade 3 or higher in severity, serious, fatal, those resulting in treatment discontinuation, and events of special interest
Change from baseline in clinical laboratory parameters | From date of randomization up to 44 months
  Percentage of participants with clinically significant laboratory results
PFS using RANO-HGG criteria | From date of randomization up to 44 months
  PFS using RANO-HGG criteria for participants with measurable contrast-enhancing disease
Corticosteroid response | From date of randomization up to 44 months
  Corticosteroid response will be measured by a confirmed 50% decrease in use of dexamethasone or equivalent
Performance status response | From date of randomization up to 44 months
  Performance status response will be measured by confirmed increase in Karnofsky Performance Status (KPS) or Lansky Performance Status (LPS)

CONTACTS AND LOCATIONS:
Locations (162):
- United States (67):
  - Banner MD Anderson Cancer Center, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA University of California Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Irvine, Orange, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Providence Saint John's Cancer Institute, Santa Monica, California
  - Stanford Cancer Center, Stanford, California
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - St Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Feinberg School of Medicine Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine - Indianapolis, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Norton Healthcare, Louisville, Kentucky
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Cancer Center - Rochester, Rochester, Minnesota
  - Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri
  - Benefis Hospital Sletten Cancer Institute, Great Falls, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Albany Medical Center, Albany, New York
  - Children's Hospital at Montefiore Medical Center, New York, New York
  - Montefiore Medical Park, New York, New York
  - Laura & Isaac Perlmutter Cancer Center - NYU ACC, New York, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Levine Cancer Institute/ Atrium Health, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Health and Services St. Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Neuro-Oncology Associates, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - UT Health Houston Neurosciences - Texas Medical Center, Houston, Texas
  - University of Texas - San Antonio - Health Science Center, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Children's Hospital of The King's Daughter, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University Of Wisconsin - Madison, Madison, Wisconsin
- FLENI Neurologia, Buenos Aires, Argentina
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Olivia Newton-John Cancer Research Institute (ONJCRI), Heidelberg, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Austria (2):
  - Medical University of Vienna - Adults, Vienna, Vienna
  - Medical University of Vienna - Pediatrics, Vienna, Vienna
- Brazil (3):
  - Hospital do GRAACC, São Paulo
  - Hcor Research Institute, São Paulo
  - Instituto Do Cancer Do Estado De São Paulo, São Paulo
- Canada (8):
  - Tom Baker Cancer Cetre, Calgary, Alberta
  - BC Cancer - The Vancouver Center, Vancouver, British Columbia
  - Children's & Women's Health Care of BC, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre Dame, Lachapelle, Montreal, Quebec
- Denmark (4):
  - Copenhagen University Hospital, Copenhagen, Capital
  - Aalborg Universitetshospital, Aalborg, North Denmark
  - F345 H.C. Andersen's Children's Hospital, Odense, Region Syddanmark
  - Odense Universitetshospital, Odense, Region Syddanmark
- Germany (11):
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - University Clinic Regensburg, Regensburg, Bavaria
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Vivantes Klinikum Neukölln, Berlin
  - Klinikum Mannheim Universitätsklinikum gGmbH, Manheim
  - Universitätsklinikum Tübingen, Tübingen
- Queen Mary Hospital, Hong Kong, Hong Kong
- Israel (7):
  - Sheba Medical Center, Ramat Gan, Tel Aviv
  - Soroka University Medical Centre, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Schneider Children's Medical Center of Israel, Petah Tikvah
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Istituto Oncologico Veneto, Padua, Veneto
- Japan (6):
  - National Cancer Center Hospital, Chūō
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyoto University Hospital, Kyoto
  - Osaka City General Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - The University of Tokyo Hospital, Tokyo
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht Cancer Center, Utrecht
- Singapore (3):
  - KK Women's and Children's Hospital, Singapore
  - National Cancer Centre, Singapore
  - National Neuroscience Institute, Singapore
- South Korea (10):
  - CHA Bundang Medical Center, Bundang-Gu, Seongnam-Si, Gyeonggido
  - Seoul National University Bundang Hospital, Bundang-gu, Seongnam-si, Gyeonggido
  - Seoul National University Hospital, Bundang-gu, Seongnam-si, Gyeonggido
  - National Cancer Center, Ilsandong-Gu, Goyang-Si, Gyeonggido
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam, Seoul Teugbyeolsi
  - Samsung Medical Center, Gangnam-Gu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Jongno-Gu, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia - Adults, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia - Pediatrics, Valencia
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Universitätsspital Zürich, Zurich
- United Kingdom (12):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Beatson West of Scotland Cancer Centre, Glasgow, Lanarkshire
  - Royal Hospital for Children (Glasgow), Glasgow, Lanarkshire
  - Clatterbridge Cancer Centre - Liverpool, Liverpool, Lancashire
  - The Christie NHS Foundation Trust, Manchester, Lancashire
  - The Royal Marsden in Sutton, Surrey, Sutton, Surrey
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - St James University Hospital, Leeds, West Yorkshire
  - The Leeds Teaching Hospitals NHS Trust, Leeds General Infimary, Leeds
  - Guy's Hospital, London
  - Churchill Hospital, Oxford